CLINICAL TRIAL: NCT06387498
Title: Testicular Tissue Cryopreservation for Fertility Preservation in Patients Facing Infertility-causing Diseases or Treatment Regimens.
Brief Title: Testicular Tissue Cryopreservation (TTC)
Acronym: TTC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-2286
Record Dates: First submitted 2022-05-13; First posted 2024-04-29 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Fertility Issues
Keywords: Fertility preservation
MeSH Terms: conditions — Infertility | interventions — Cryopreservation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Testicular Tissue Cryopreservation (Experimental): Enrolled participants will undergo a testicular tissue biopsy. The method and amount of tissue procurement will be at the discretion of the surgeon.
  Interventions: Procedure: Testicular tissue biopsy and cryopreservation

INTERVENTIONS:
Procedure: Testicular tissue biopsy and cryopreservation — Surgical Procurement of Testicular Tissue: At early stages of technology development, simple orchiectomy (removal of one entire testicle) may give the best chance of preserving sufficient cells for effective therapy. However, incisional biopsy of up to 25% of tissue from one testis (wedge resection) will also be presented to the patient as an alternative option. The amount of testicular parenchyma removed will be at the discretion of the surgeon.

SUMMARY:
The "Testicular Tissue Cryopreservation" study is open to a subset of patients facing disease or treatment regimens that could lead to infertility (gonadotoxic therapies). For some of these patients, experimental testicular tissue cryopreservation is the only fertility preservation option available. The overall objective of this study is to determine the feasibility and acceptability of testicular tissue cryopreservation in male patients of all ages who have a condition or will undergo a treatment that can cause infertility.

DETAILED DESCRIPTION:
For male patients who currently have no options for fertility preservation, this research proposal will enable optimization of testicular tissue procurement and processing, cryopreservation, and diagnosis/elimination of malignant cell contamination to ensure safety for future fertility-restoring treatments. While results from animal models and human organ donor experiments support the efficacy of testicular tissue/cell cryopreservation for fertility preservation and subsequent restoration, rigorous safety and efficacy data in human patients who will undergo infertility-causing therapies is lacking. However, the patients being recruited for this study currently have no options for future therapies aimed at fertility preservation without the preservation of their testicular tissue/cells prior to treatment. Thus, the current study will provide a potential resource for future fertility restoration.

ELIGIBILITY:
Inclusion Criteria:

1. Male at any age.
2. Scheduled to undergo surgery, chemotherapy, drug treatment and/or radiation for the treatment or prevention of a medical condition or malignancy with risk of causing permanent and complete loss of subsequent testicular function. Be in significant risk of infertility as defined by:

   * Cyclophosphamide equivalent dose (CED) ≥4 g/m2
   * Total body irradiation (TBI)
   * Testicular radiation >2.5 Gy
   * Cisplatin 500 mg/m2
   * Bone Marrow Transplant (BMT)
3. Or have a medical condition or malignancy that requires removal of all or part of one or both testicles.
4. Or have newly diagnosed or recurrent disease. Those who were not enrolled at the time of initial diagnosis (i.e., patients with recurrent disease) are eligible if they have not previously received therapy that is viewed as likely to result in complete and permanent loss of testicular function.
5. Have two testicles if undergoing elective removal of a testicle for fertility preservation only. Note: removal of both testicles will limit fertility preservation options.
6. Sign an approved informed consent and authorization permitting the release of personal health information. The patient and/or the patient's legally authorized guardian must acknowledge in writing that consent for specimen collection has been obtained, in accordance with institutional policies approved by the U.S. Department of Health and Human Services.
7. Consent for serum tests for infectious diseases [including Hepatitis B Surface Antigen, Hepatitis C Virus (HCV) Antibody, and Human Immunodeficiency Virus (HIV) antigen/antibody screen to be performed at the time of testicular tissue harvesting.
8. Undergo a full history and physical examination and obtain standard pre-operative clearance (based on the most recent American College of Cardiology/American Heart Association (ACC/AHA) Guideline for Perioperative Cardiovascular Evaluation for Noncardiac Surgery) as determined by their primary surgeon.

Exclusion Criteria

Patients will be ineligible for participation in this study if they are:

1. Diagnosed with psychological, psychiatric, or other conditions which prevent giving fully informed consent.
2. Diagnosed with an underlying medical condition that significantly increases their risk of complications from anesthesia and surgery.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility, as Assessed via the Percentage of Eligible Patients who do a Procedure | Up 3 months after prescribed gonadotoxic therapy
  Determine feasibility of testicular tissue cryopreservation (TTC) in male patients receiving gonadotoxic therapies who desire fertility preservation. Calculated by the percentage of eligible patients that elect to proceed with TTC.
Feasibility, as Assessed via Percentage of Patients who Attempted a Procedure who were able to Cryopreserve | Up to 48 hours after testicular tissue biopsy
  Determine feasibility of testicular tissue cryopreservation (TTC) in male patients receiving gonadotoxic therapies who desire fertility preservation. Calculated by the number of study participants whose tissue was successfully cryopreserved.
Safety, as Assessed via the Number of Participants with At Least One Pre-specified Adverse Event | Every six months throughout the life of the study (up to 7 years)
  The investigators will determine the safety of testicular tissue cryopreservation (TTC) in male patients receiving gonadotoxic therapies who desire fertility preservation. The number of participants with at least one of the following adverse events: 1) Bleeding, 2) Post-op infection, or 3) Long-term pain.
Safety, as Assessed via the Number of Participants with At Least One Pre-specified Adverse Event | 24 hours of the procedure
  The investigators will determine the safety of testicular tissue cryopreservation (TTC) in male patients receiving gonadotoxic therapies who desire fertility preservation. The number of participants with bleeding.
Safety, as Assessed via the Number of Participants with At Least One Pre-specified | within 72 hours of the procedure
  The investigators will determine the safety of testicular tissue cryopreservation (TTC) in male patients receiving gonadotoxic therapies who desire fertility preservation. The number of participants with post-op infection.
Safety, as Assessed via the Number of Participants with At Least One Pre-specified | Assessed at 6 months
  The investigators will determine the safety of testicular tissue cryopreservation (TTC) in male patients receiving gonadotoxic therapies who desire fertility preservation. The number of participants with long-term pain.

SECONDARY OUTCOMES:
Acceptability, as Assessed via Annual Survey Regret Score | Annually until the age of majority for the male participant
  The Decision Regret Scale measures distress or remorse after a health care decision. Possible scores range from 0-100, with higher scores indicating high regret.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Corkum, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No